CLINICAL TRIAL: NCT04247880
Title: Advancing Women in the Sheet Metal Workers' Trade: A Coordinated Mentoring Program to Promote Safety, Health, and Well-being
Brief Title: The Use of Mentoring to Promote Well-being for Female SMART Members
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The Center for Construction Research and Training (CPWR) (Unknown); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marissa Baker, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00009270; U60OH009762-11 (NIH)
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Harassment, Non-Sexual; Harassment, Sexual; Bullying, Workplace; Mental Stress; Work-Related Condition; Work-related Injury; Work Related Stress
MeSH Terms: conditions — Harassment, Non-Sexual; Sexual Harassment; Occupational Stress; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentees (Experimental): This arm consists of apprentice-level, female-identifying construction workers who will receive active mentorship (the intervention) for two years from trained journey-level mentors.
  Interventions: Behavioral: Mentoring program
- Control Apprentices (No Intervention): This arm consists of apprentice-level, female-identifying construction workers who will not receive mentorship.

INTERVENTIONS:
Behavioral: Mentoring program — Apprentice-level female construction workers will be assigned to a mentor who has gone through a rigorous mentorship training. Participants will be asked to meet with a mentor at least 4 times/year in person to discuss the challenges of being a female in construction, learn coping mechanisms, and otherwise discuss the unique challenges of the job environment.
  Arms: Mentees

SUMMARY:
Women are highly underrepresented in the construction skilled trades. In addition to facing the industry's well-known physical risks, women are subjected to discrimination, harassment, and skills under-utilization. As a result, tradeswomen have increased risk for injury, stress-related health effects, and high attrition rates from apprenticeship programs, thus perpetuating their minority status. Mentoring is a well-established technique for learning technical and personal navigation skills in new or challenging social environments. The investigators propose development and dissemination of a mentorship program through local unions of the International Association of Sheet Metal, Air, Rail and Transportation Workers (SMART), and evaluating its success in reducing women's injury and work stress, while improving retention.

DETAILED DESCRIPTION:
Journey-level workers will be trained on effective mentoring techniques, and matched to approximately 100 women apprentices within participating local unions. Mentees will be followed for two years within the mentorship program, with another 100 women apprentices in locals not receiving the mentorship training similarly followed as controls. The impact of participation in mentoring programs will be measured through apprentices' experience of stress, coping mechanisms, safety climate, and retention in the apprenticeship programs. Specifically, the investigators propose to:

Aim 1: Develop a mentorship training program for journey-level sheet metal workers to assist women apprentices in navigating the challenges faced by women in trades

Aim 2: Disseminate the training and assist locals in developing effective mentorship programs

Aim 3: Evaluate the effectiveness of the mentoring programs specified in Aims 1 and 2

Aim 4: Disseminate the best practices for supporting women apprentices in the skilled trades.

ELIGIBILITY:
Inclusion Criteria:

* All mentors must be journey-level sheet metal workers that are members of the SMART (International Association of Sheet Metal, Air, Rail, and Transportation Workers) Union. All mentees and control apprentices must be apprentice-level sheet metal workers that are members of the SMART Union, and identify as woman.

Exclusion Criteria:

* No exclusions will be made on the basis of sex, race, ethnicity, age, disability or religion for mentors, mentees, and control apprentices. No exclusions will be made on the basis of gender for mentors. For mentees and control apprentices, those that do not identify as a woman will be excluded.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mentors can be both male- and female-identifying. Mentees and control apprentices will be all female-identifying.
Enrollment: 96 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marissa G Baker, PhD, Principal Investigator — University of Washington; Lily M Monsey, BA, Study Director — University of Washington
Locations (19):
- United States (19):
  - Phoenix Area Local 359, Phoenix, Arizona
  - Sheet Metal Workers Local 105, Glendora, California
  - Sheet Metal Workers Local 104, San Jose, California
  - Sheet Metal Workers Local 9, Denver, Colorado
  - Sheet Metal Workers Local 85, Atlanta, Georgia
  - Hawaii Sheet Metal Workers Local 293, Honolulu, Hawaii
  - Sheet Metal Workers Local 73, Hillside, Illinois
  - Sheet Metal Workers Local 20, Indianapolis, Indiana
  - Sheet Metal Workers Local 17, Dorchester, Massachusetts
  - Sheet Metal Workers Local 63, Springfield, Massachusetts
  - Sheet Metal Workers Local 10, Maplewood, Minnesota
  - Sheet Metal Workers Local 36, St Louis, Missouri
  - Sheet Metal Workers Local 49, Albuquerque, New Mexico
  - Sheet Metal Workers Local 28, New York, New York
  - Columbus Sheet Metal Workers Apprenticeship, Columbus, Ohio
  - Sheet Metal Workers Local 16, Portland, Oregon
  - Sheet Metal Workers Local 19, Philadelphia, Pennsylvania
  - Sheet Metal Workers Local 67, San Antonio, Texas
  - Sheet Metal Workers Local Union 66, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details Recruitment for round 1 of the study took place from March-May 2021. Recruitment for round 2 of the study took place from July-December 2023. All recruitment activity took place remotely via video conferencing software, email and phone, with union locals as the recruitment locations.
Pre-assignment Details: Evolving impacts of the COVID-19 pandemic influenced the environmental conditions between the period of participant enrollment and the time participants were assigned to each arm. No enrolled participants were excluded from the study before assignment.
Groups:
- Mentees: Mentees were assigned to trained mentors to support them with informational, appraisal, and tangible social support through development of active listening, goal setting, problem solving, and self advocacy skills.
- Control Apprentices: Control apprentices were not assigned to a trained mentor during the study period.
Period: Overall Study
Arm/Group | Mentees | Control Apprentices
Started | 56 | 40
Completed | 29 | 23
Not Completed | 27 | 17
Not completed — Lost to Follow-up | 24 | 17
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: 51 and 39 mentees and apprentices, respectively, completed the baseline measures in the survey. For job satisfaction and social support, all records are reported in the data table. In the case of perceived stress, 48 records for mentees and 38 records for controls are reported in the data table. The reason for this is because not all participants responded to all questions pertaining to perceived stress, so we could not analyze all records for this outcome.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mentees | Control Apprentices | Total
Number analyzed (Participants) | 51 | 39 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 39 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 28 [18 to 45] | 27 [18 to 46] | 28 [18 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 39 | 90
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 26 | 54
  Black or African American | 5 | 8 | 13
  Hispanic, Latinx, or Spanish Origin | 6 | 4 | 10
  Other | 12 | 1 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 39 | 88
  Canada | 2 | 0 | 2
Perceived Stress [Mean (Standard Deviation); unit: units on a scale] — Measures of feelings of stress among the female workers from the Perceived Stress Scale (PSS) where higher scores indicate a worse outcome. Minimum value is 0 and maximum value is 40. Population: Numbers in each row differ because not all participants answered all questions pertaining to percieved stress on the baseline measure.
  units on a scale
    number analyzed (Participants) | 48 | 38 | 86
    (all) | 18.1 (8.1) | 14.1 (7.4) | 16.3 (7.8)
Social Support [Mean (Standard Deviation); unit: units on a scale] — Measures of social support both in and out of work from MOS (Medical Outcomes Study) Social Support Survey. Higher scores indicate greater feelings of social support. Minimum value of 1 and maximum value of 5.
  units on a scale | 4.4 (0.7) | 4.4 (0.6) | 4.4 (0.7)
Job Satisfaction [Mean (Standard Deviation); unit: units on a scale] — Measures of job satisfaction from the Job Satisfaction Survey (JSS) where higher scores indicate higher job satisfaction. Minimum value is 1 and maximum value is 6.
  units on a scale | 3.1 (0.5) | 3.1 (0.6) | 3.1 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Stress
Description: Measures of feelings of stress among the female workers from the Perceived Stress Scale (PSS) where higher scores indicate a worse outcome. Minimum value is 0 and maximum value is 40.
Time Frame: 1 year period
Population: Mentees and control apprentices who completed all questions on the end-of-year survey pertaining to perceived stress
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mentees | Control Apprentices
Number analyzed (Participants) | 19 | 20
score on a scale | 17.6 (6.5) | 13.1 (4.5)

2. Primary Outcome: Job Satisfaction
Description: Measures of job satisfaction from the Job Satisfaction Survey (JSS) where higher scores indicate higher job satisfaction. Minimum value is 1 and maximum value is 6.
Time Frame: 1 year period
Population: participants who completed or partially competed the baseline survey, including questions pertaining to this measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mentees | Control Apprentices
Number analyzed (Participants) | 19 | 20
score on a scale | 2.9 (0.6) | 3.0 (0.4)

3. Primary Outcome: Social Support
Description: Measures of social support both in and out of work from the Medical Outcomes Study (MOS) Social Support Survey. Higher scores indicate greater feelings of social support. Minimum value of 1 and maximum value of 5.
Time Frame: 1 year period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mentees | Control Apprentices
Number analyzed (Participants) | 19 | 21
score on a scale | 4.4 (0.9) | 4.3 (0.8)

ADVERSE EVENTS:
Time Frame: Adverse events were not assessed as they were not applicable to our study.
Description: We were not collecting data on typical adverse events such as death, injury, unexpected reactions due to the mentorship program because this was not applicable to our study.
Arm/Group | Mentees | Control Apprentices
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
COVID-19 impacted the delivery and uptake of the intervention, as well as our ability to recruit and retain participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT04247880/Prot_SAP_ICF_000.pdf